CLINICAL TRIAL: NCT02199977
Title: Innovative Public-private Partnership to Target Subsidized Antimalarials in the Retail Sector
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Moi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00052602; 1R01AI110478-01 (NIH)
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Fever; Malaria
Keywords: Malaria; Antimalarial subsidy; Malaria rapid diagnostic test (RDT); public-private partnership
MeSH Terms: conditions — Fever; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- test only (free) (Other): The participant is entitled to a free malaria rapid diagnostic test, but no ACT voucher.
  Interventions: Other: Free Malaria Rapid Diagnostic Test
- test (free) & conditional ACT voucher (Other): The participant is entitled to a free malaria rapid diagnostic test, and an ACT voucher conditional on a positive test result.
  Interventions: Other: Free Malaria Rapid Diagnostic Test; Other: Conditional ACT voucher
- test only (not free) (Other): The participant is entitled to a malaria rapid diagnostic test for a charge (i.e., not for free), but no ACT voucher.
  Interventions: Other: Malaria Rapid Diagnostic test for a charge
- test (not free) & conditional ACT voucher (Other): The participant is entitled to a malaria rapid diagnostic test for a charge (i.e., not for free), and an ACT voucher conditional on a positive test result.
  Interventions: Other: Conditional ACT voucher; Other: Malaria Rapid Diagnostic test for a charge

INTERVENTIONS:
Other: Free Malaria Rapid Diagnostic Test — Malaria RDT is offered free if patients choose to be tested
  Arms: test (free) & conditional ACT voucher; test only (free)
Other: Conditional ACT voucher — Participants will be eligible to receive a drug subsidy for a set amount (in the form of a voucher) conditional on a positive malaria test. When a conditional subsidy is offered, it is valid for use on a "Green Leaf" approved malaria drug.
  Arms: test (free) & conditional ACT voucher; test (not free) & conditional ACT voucher
Other: Malaria Rapid Diagnostic test for a charge — Participants can receive a malaria RDT for a set amount (i.e., not for free).
  Arms: test (not free) & conditional ACT voucher; test only (not free)

SUMMARY:
There are compelling medical and public health reasons to reduce unnecessary consumption of antimalarials and strong evidence to support the use of RDTs in malaria case management. The primary study hypothesis to be tested is that clients who know they will receive a subsidy conditional on a positive test are more likely to opt for testing before deciding which drug to buy. The primary endpoint is whether subjects choose to be tested for malaria with a rapid diagnostic test. The secondary endpoint is whether they purchased an artemisinin combination therapy (ACT) or not. The primary outcome of interest is to compare the proportion of participants who choose to receive a free malaria diagnostic test when they can receive a subsidy for a discounted drug conditional on a positive test (Group A compared to Group B) compared to those without the offer of a conditional subsidy. The investigators will use an experimental design that randomly assigns clients to one of four groups. Field workers will canvas households in the study area looking for individuals who have fever or history of fever or illness in the last 24 hours (current illness) who have not yet taken drugs or sought treatment outside the home. Clients who meet the inclusion criteria and give verbal consent to participate will be randomly assigned to one of the four groups. They will be given the location and contact information for their local community health worker who can provide a malaria rapid diagnostic test if they choose to be tested. They will also complete a survey tool. One week later, the field worker will return to interview the participant and determine whether they were tested, what action they took for their illness, what medicine they purchased and how much they paid. The investigators will summarize clients' choice by the four randomized study groups.

ELIGIBILITY:
Inclusion Criteria:

* Client is older than 1 year
* Client has fever or history of fever or feeling unwell with a malaria-like illness within the last 24 hours
* Client or their parent/legal guardian consents to participate

Exclusion Criteria:

* Client has signs of severe disease or other problem requiring immediate referral to a community health worker (CHW) / health facility
* Client has already sought treatment, purchased medicine or taken medicine for the current illness.

Note:

If more than one febrile person who meet the inclusion criteria are found in a single household, all of the individuals will be enrolled in the same group, but only one individual (the first enrolled) will be used for the purposes of the analysis.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Effect of conditional drug subsidy on proportion of participants who choose to receive a free malaria diagnostic test | Within two days of group assignment
  The primary outcome of interest is to compare the proportion of participants who choose to receive a free malaria diagnostic test when they can receive a subsidy for a discounted drug conditional on a positive test compared to those without the offer of a conditional subsidy.

SECONDARY OUTCOMES:
Effect of malaria RDT subsidy on the uptake of testing (free versus paid RDT) | Within 2 days of group assignment
Effect of a conditional ACT subsidy on uptake of testing when the RDT is not free. | Within 2 days of group assignment

OTHER OUTCOMES:
Percent of clients with a negative test, a positive test or no test who choose to purchase an ACT in all four groups. | Within 2 days of test results

CONTACTS AND LOCATIONS:
Overall Officials: Wendy O'Meara, PhD, Principal Investigator — Duke University
Locations (1):
- Moi University, Eldoret, Kenya

REFERENCES:
- [Derived] Prudhomme O'Meara W, Mohanan M, Laktabai J, Lesser A, Platt A, Maffioli E, Turner EL, Menya D. Assessing the independent and combined effects of subsidies for antimalarials and rapid diagnostic testing on fever management decisions in the retail sector: results from a factorial randomised trial in western Kenya. BMJ Glob Health. 2016 Sep 28;1(2):e000101. doi: 10.1136/bmjgh-2016-000101. eCollection 2016. PMID 28588946